CLINICAL TRIAL: NCT05824260
Title: Risk Factors for Postoperative Complications in Major Non-cardiac Surgery: Post-hoc Analysis of the OPHIQUE Multicentre Study
Acronym: MULTIPAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2022_843_0099
Record Dates: First submitted 2023-03-28; First posted 2023-04-21 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-03

CONDITIONS: Goal Directed Therapy; Postoperative Morbidity; Individualised Target; Postopera Mortality
Keywords: Goal directed therapy; postoperative morbi-mortality; individualised target

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with complications
- patients without complication

SUMMARY:
Post-operative morbidity and mortality is related to many factors related to the patient's condition, the intra-operative period and the optimisation of intra-operative haemodynamic and respiratory parameters. Many studies have looked at the determinants and factors that increase postoperative complications. However, these have been randomised studies looking at one parameter in particular.

This analysis would be the first to investigate the determinants of postoperative complications in a large population of patients undergoing major non-cardiac surgery. This is a post-hoc analysis of patients included in the OPHIQUE study, whose main objective was to evaluate intraoperative haemodynamic management guided by a marker of tissue hypoperfusion (the respiratory quotient).

ELIGIBILITY:
Inclusion Criteria:

* Abdominal, orthopaedic or vascular surgery under general anaesthesia and with an estimated duration of surgery > 2 hours
* Adult patients (age ≥ 18 years)
* ASA score ≥ II
* Patient with at least two of the following comorbidities: age > 50 years, high blood pressure (HTA), heart failure, ECG abnormality, smoking, stroke, transient ischemic attack (TIA), peripheral arterial disease (PAD), insulin-dependent or non-insulin-dependent diabetes mellitus (NIDDM), ascites, chronic renal failure (CRF)
* Signature of the consent form
* Affiliation to a social security scheme

Exclusion Criteria:

* Severe untreated or unbalanced hypertension
* Preoperative renal failure on dialysis
* Acute heart failure
* Acute coronary insufficiency
* Vascular surgery with renal plasty
* Cardiac surgery
* Permanent laparoscopy
* Chronic respiratory failure with home oxygen therapy
* Acute respiratory distress syndrome with FiO2>60%.
* Preoperative shock
* Surgery under spinal anaesthesia and epidural only
* Refusal to participate by the patient
* Pregnant, parturient or breastfeeding women
* Patients under guardianship or curators, under court protection or deprived of public rights
* The patient already included in another therapeutic trial with an experimental molecule
* Emergency surgery
* Patients who do not want their personal data to be used in the framework of the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Abdominal, orthopaedic or vascular surgery under general anaesthesia and with an estimated duration of surgery > 2 hours
  * Adult patients (age ≥ 18 years)
  * ASA score ≥ II
  * Patient with at least two of the following comorbidities: age > 50 years, high blood pressure (HTA), heart failure, ECG abnormality, smoking, stroke, transient ischemic attack (TIA), peripheral arterial disease (PAD), insulin-dependent or non-insulin-dependent diabetes mellitus (NIDDM), ascites, chronic renal failure (CRF)
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
NUmber of risk factors associated with postoperative morbidity in major non-cardiac surgery | 2 years
Number of risk factors associated with postoperative mortality in major non-cardiac surgery | 2 years

SECONDARY OUTCOMES:
Number of risk factors associated with the occurrence of postoperative renal dysfunction. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No